CLINICAL TRIAL: NCT05357040
Title: Evaluation of the Antidepressant Effects of Nitrous Oxide in People With Major Depressive Disorder
Brief Title: Antidepressant Effects of Nitrous Oxide
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: The Alfred (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB18-1856
Record Dates: First submitted 2021-11-09; First posted 2022-05-02 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression
Keywords: Depression; Antidepressant; Nitrous Oxide
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression | interventions — Endothelium-Dependent Relaxing Factors; Inhalation; Nitrous Oxide

STUDY DESIGN:
Intervention Model Description: Parallel-group, controlled trial; randomized participants (1:1) to nitrous oxide (Nitrous group) or oxygen-air mixture (FiO2 ≈0.3, Control group). The Nitrous group will be further randomly assigned to either 50% nitrous oxide in oxygen (FiO2 0.5) or 25% nitrous oxide in oxygen (FiO2 0.75).
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient and assessor blinded to study group assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment; Nitrous Oxide 50% or 25%, group (Active Comparator): Four-weekly, 60-minute inhalation sessions of 25% or 50% nitrous oxide, randomly assigned.
  Interventions: Drug: Nitrous oxide gas for inhalation
- Control; Oxygen-air mixture, group (Placebo Comparator): Four-weekly, 60-minute inhalation sessions of an oxygen and air mixture.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitrous oxide gas for inhalation — 60-minute sessions of inhaled 50% nitrous oxide in oxygen (FiO2 0.5) or 25% nitrous oxide in oxygen (FiO2 0.75), administered weekly for 4-weeks.
  Administration will be under the direct supervision of a licensed practitioner who is experienced in the use and administration of the study drug, and is familiar with the indications, effects, dosages, methods, and frequency and duration of administration, and with the hazards, contraindications, and side effects and the precautions to be taken (MD, or CRNA); with study patient monitoring of pulse oximetry, heart rate, respiratory, non-invasive blood pressure, and end-tidal carbon dioxide.
  Other Names: N2O; Laughing gas; Nitrous Oxide; Nitrous
  Arms: Treatment; Nitrous Oxide 50% or 25%, group
Drug: Placebo — 60-minute sessions of inhaled oxygen-air mixture (FiO2 ≈0.3) to be administered weekly for 4-weeks.
  Administration will be under the direct supervision of a licensed practitioner who is experienced in the use and administration of the study drug, and is familiar with the indications, effects, dosages, methods, and frequency and duration of administration, and with the hazards, contraindications, and side effects and the precautions to be taken (MD, or CRNA); with study patient monitoring of pulse oximetry, heart rate, respiratory, non-invasive blood pressure, and end-tidal carbon dioxide.
  Arms: Control; Oxygen-air mixture, group

SUMMARY:
To evaluate the acute and sustained antidepressant effects of nitrous oxide in people with major depressive disorder; and further evaluate these effects by identifying the optimal dose and regimen to guide current practice, and to plan a future large pragmatic trial.

DETAILED DESCRIPTION:
The investigators are conducting a randomized controlled trial to evaluate the antidepressant effects of nitrous oxide in people with Major Depressive Disorder (MDD). MDD is a global medical condition that causes significant health and economic burden. Recent studies have shown that a single dose of ketamine, an NMDA-antagonist, has fast and long lasting anti-depressant effect. Nitrous oxide, another NMDA-antagonist, is widely used for anesthesia and analgesia, safer to administer and has fewer side effects than ketamine.

A randomized controlled crossover feasibility study showed significant reduction in depressive symptoms at 2 and 24 hours after a single 1-hour treatment session of inhaled nitrous oxide compared with placebo. Nitrous oxide is inexpensive and can be safely administered by any trained clinician. If found to be efficacious, it could be used to provide rapid anti-depressant effect whilst the benefit of traditional anti-depressants has its delayed effect. Another potential application could be in acutely suicidal patients.

This trial will enable confirmation and extension of the findings from the feasibility study, and identify the optimal dose and regimen in a broader population of those with MDD. Participants will be randomized to receive a weekly 1-hour inhalational session of either nitrous oxide or placebo (oxygen-air mixture) for 4 weeks, and the nitrous group will be further randomly assigned to a dose of 50% or 25% nitrous oxide. Depression severity and outcomes related to treatment responses will be continuously assessed by a 'blinded-to-randomization' psychiatry (MD) rater at weekly intervals during study patient participation, using validated psychiatric diagnostics (Hamilton Depression Rating Scale-21 [HDRS-21 or HAM-D]; Profile of Mood States [POMS]; Computerized Adaptive Test-Mental Health [CAT-MH]; Sheehan-STS [S-STS]; Visual Analog Scale [VAS]).

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years, both sexes)
2. DSM-5 criteria for MDD without psychosis, as determined using a structured clinical interview [Mini International Neuropsychiatric Interview], MDD, defined by a pre-treatment score >16 on the HDRS-21 scale and meeting DSM-5 for MDD

Exclusion Criteria:

1. A current or past history of bipolar disorder, schizophrenia, or schizoaffective disorder.
2. Current obsessive-compulsive disorder, panic disorder, or documented Axis II diagnoses
3. Active suicidal intention, as determined by clinical interview assessment tool (Sheehan-STS) and clinical examination
4. Active or recent (<12 months) substance use disorder; excluding nicotine
5. Administration of NMDA-antagonists (e.g., ketamine) in previous 3 months
6. Ongoing treatment with ECT
7. Presence of acute medical illness that could interfere with study participation, including significant pulmonary disease
8. Pregnancy or breastfeeding
9. Any contraindications to the use of nitrous oxide (e.g., pneumothorax, middle ear occlusion, elevated intracranial pressure, chronic cobalamin or folate deficiency unless treated with folic acid or vitamin B12).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in HDRS-21 score | Over 4-weeks from baseline
  Monitor changes in Hamilton Depression Rating Scale-21 (HDRS-21) scores to determine whether a series of four, 60-minute sessions of inhaled nitrous oxide vs placebo (once-per-week) has significant antidepressant activity.
  The HDRS-21 is an interview-based psychiatric diagnostic used to evaluate depression severity. Scores are calculated by using the first 17 responses of this 21 item questionnaire.
  Higher scores are associated with more severe depression:
  0 - 7 = Normal 8 - 13 = Mild Depression 14-18 = Moderate Depression 19 - 22 = Severe Depression > 23 = Very Severe Depression Max score = 52

SECONDARY OUTCOMES:
Treatment response | At 24-hours (following treatment-1)
  Treatment response (≥50% reduction on HDRS-21) to nitrous oxide vs placebo will be measured.
Changes in 'Profile of Mood States' scores | Up to 1-week (following treatment-1)
  Monitoring daily mood changes using the Profile of Mood States (POMS) a validated 'self-report' psychological diagnostic containing 65 emotions or 'mood states' to determine the pattern of treatment response
  Patients rank their current mood states using a scale of 'not-at-all', 'a-little', 'moderately', 'quite-a-lot', 'extremely'. Responses are scored to calculated the Total Mood Disturbance (TMD):
  TMD = (tension + depression + anger + fatigue + confusion) - Vigor
Sustainability of treatment response | Over 7-weeks (length of study participation).
  Determine sustained response and remission following study treatments (nitrous vs placebo) using Hamilton Depression Rating Scale-21 (HDRS-21) score.
  The HDRS-21 is an interview-based psychiatric diagnostic used to evaluate depression severity. Scores are calculated by using the first 17 responses of this 21 item questionnaire.
  Higher scores are associated with more severe depression:
  0 - 7 = Normal 8 - 13 = Mild Depression 14-18 = Moderate Depression 19 - 22 = Severe Depression > 23 = Very Severe Depression Max score = 52
Treatment dose response comparison | Over 7-weeks (length of study participation)
  Compare dose response of 25% vs 50% nitrous oxide to establish whether the concentration is related to outcome.
  Determined with treatment-by-dose (group) interaction term in a logistic regression model to assess for statistical significance.
Treatment cycle compliance | Over 4-weeks (weekly treatment sessions)
  Evaluate compliance to complete 4-cycle inhalation treatments of nitrous oxide vs placebo.
  Determined by ability, inability, or refusal to receive all 4-treatments of randomized inhalation sessions (nitrous oxide vs placebo).
Changes in Computerize Adaptive Testing - Mental Health (CAT-MH) 'depression' scores | Over 7-weeks (length of study participation) from Baseline
  This CAT-MH is a validated self-reporting diagnostic that adaptively selects a small optimal set of items from a large bank of approximately 1,500 items, targeted to individuals current or historical level of severity and likelihood of 'depression'.
  Generated scores include severity and liklihood percentile:
  - depression = (%) normal, mild, moderate, severe
Changes in Computerize Adaptive Testing - Mental Health (CAT-MH) 'anxiety' scores | Over 7-weeks (length of study participation) from Baseline
  This CAT-MH is a validated self-reporting diagnostic that adaptively selects a small optimal set of items from a large bank of approximately 1,500 items, targeted to individuals current or historical level of severity and likelihood of 'anxiety'.
  Generated scores include severity and liklihood percentile:
  - anxiety = (%) normal, mild, moderate, severe
Changes in Computerize Adaptive Testing - Mental Health (CAT-MH) 'suicide' scores | Over 7-weeks (length of study participation) from Baseline
  This CAT-MH is a validated self-reporting diagnostic that adaptively selects a small optimal set of items from a large bank of approximately 1,500 items, targeted to individuals current or historical level of severity and likelihood of 'suicide'.
  Generated scores include severity and liklihood percentile:
  - suicide = (%) low, intermediate, high
Suicidal ideation tracking | Over 7-weeks (length of study participation) from Baseline
  Suicidal ideation will be be tracked using the Sheehan Suicidality Tracking Scale (S-STS), a validated self-report diagnostic tool designed to assess and monitor suicidality.
  The standard S-STS consists of 14 core questions related to suicidality phenomena and is designed for use in clinical research studies and in clinical settings.
  Scores are summed based on individual responses 'not-at-all = 0', 'a little = 1', 'moderately = 2', 'very = 3', 'extremely = 4', to generate a summated score (total score), individual factor scores for suicidal ideation, suicidal intent, suicidal planning, suicidal behavior, and non-suicidal self-injury.
  All results are monitored in real time by a trained psychiatry (MD) rater.
Visual Analog Scale (VAS) | At Baseline (Prior to treatment-1)
  The VAS is a unidimensional measure of pain intensity and use in the field of psychology to measure 'well-being'.
  Patients mark on a line the point that they feel represents their perception of their current state, with the score determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.
  The range of score from 0-100 mm and represent: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Treatment remission | At 24-hours (following treatment-1)
  Treatment remission (HDRS-21 ≤7 points) to nitrous oxide vs. placebo will be measured.

OTHER OUTCOMES:
Adverse Events | Over 7-weeks (length of study participation).
  Psychiatric AEs, such as new suicidal ideation and psychotic symptoms; AEs such as nausea and vomiting; or any other AEs determined probably, possibly, or unrelated to the study intervention.
  Study patient safety is monitored by the investigators (MD) with experience in critical care anesthesia, and psychiatry, as well as an experienced clinical research team responsible for monitoring and reporting events.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nagele, MD, MSc, Principal Investigator — University of Chicago, Department of Anesthesia and Critical Care; Paul Myles, MD, Principal Investigator — The Alfred Hospital, Department of Anesthesiology and Perioperative Medicine
Locations (2):
- University of Chicago Medicine, Chicago, Illinois, United States
- The Alfred Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] Conway CR, George MS, Sackeim HA. Toward an Evidence-Based, Operational Definition of Treatment-Resistant Depression: When Enough Is Enough. JAMA Psychiatry. 2017 Jan 1;74(1):9-10. doi: 10.1001/jamapsychiatry.2016.2586. No abstract available. PMID 27784055
- [Background] McIntyre RS, Filteau MJ, Martin L, Patry S, Carvalho A, Cha DS, Barakat M, Miguelez M. Treatment-resistant depression: definitions, review of the evidence, and algorithmic approach. J Affect Disord. 2014 Mar;156:1-7. doi: 10.1016/j.jad.2013.10.043. Epub 2013 Nov 15. PMID 24314926
- [Background] Schlaepfer TE, Agren H, Monteleone P, Gasto C, Pitchot W, Rouillon F, Nutt DJ, Kasper S. The hidden third: improving outcome in treatment-resistant depression. J Psychopharmacol. 2012 May;26(5):587-602. doi: 10.1177/0269881111431748. Epub 2012 Jan 11. PMID 22236505
- [Background] Sackeim HA. The definition and meaning of treatment-resistant depression. J Clin Psychiatry. 2001;62 Suppl 16:10-7. PMID 11480879
- [Background] Kim YK, Na KS. Role of glutamate receptors and glial cells in the pathophysiology of treatment-resistant depression. Prog Neuropsychopharmacol Biol Psychiatry. 2016 Oct 3;70:117-26. doi: 10.1016/j.pnpbp.2016.03.009. Epub 2016 Apr 1. PMID 27046518
- [Background] Lener MS, Niciu MJ, Ballard ED, Park M, Park LT, Nugent AC, Zarate CA Jr. Glutamate and Gamma-Aminobutyric Acid Systems in the Pathophysiology of Major Depression and Antidepressant Response to Ketamine. Biol Psychiatry. 2017 May 15;81(10):886-897. doi: 10.1016/j.biopsych.2016.05.005. Epub 2016 May 12. PMID 27449797
- [Background] Palucha-Poniewiera A, Pilc A. Glutamate-Based Drug Discovery for Novel Antidepressants. Expert Opin Drug Discov. 2016 Sep;11(9):873-83. doi: 10.1080/17460441.2016.1213234. Epub 2016 Aug 2. PMID 27409299
- [Background] Gerhard DM, Wohleb ES, Duman RS. Emerging treatment mechanisms for depression: focus on glutamate and synaptic plasticity. Drug Discov Today. 2016 Mar;21(3):454-64. doi: 10.1016/j.drudis.2016.01.016. Epub 2016 Feb 6. PMID 26854424
- [Background] Autry AE, Adachi M, Nosyreva E, Na ES, Los MF, Cheng PF, Kavalali ET, Monteggia LM. NMDA receptor blockade at rest triggers rapid behavioural antidepressant responses. Nature. 2011 Jun 15;475(7354):91-5. doi: 10.1038/nature10130. PMID 21677641
- [Background] McCloud TL, Caddy C, Jochim J, Rendell JM, Diamond PR, Shuttleworth C, Brett D, Amit BH, McShane R, Hamadi L, Hawton K, Cipriani A. Ketamine and other glutamate receptor modulators for depression in bipolar disorder in adults. Cochrane Database Syst Rev. 2015 Sep 29;(9):CD011611. doi: 10.1002/14651858.CD011611.pub2. PMID 26415966
- [Background] Katalinic N, Lai R, Somogyi A, Mitchell PB, Glue P, Loo CK. Ketamine as a new treatment for depression: a review of its efficacy and adverse effects. Aust N Z J Psychiatry. 2013 Aug;47(8):710-27. doi: 10.1177/0004867413486842. Epub 2013 May 9. PMID 23661785
- [Background] Hu YD, Xiang YT, Fang JX, Zu S, Sha S, Shi H, Ungvari GS, Correll CU, Chiu HF, Xue Y, Tian TF, Wu AS, Ma X, Wang G. Single i.v. ketamine augmentation of newly initiated escitalopram for major depression: results from a randomized, placebo-controlled 4-week study. Psychol Med. 2016 Feb;46(3):623-35. doi: 10.1017/S0033291715002159. Epub 2015 Oct 19. PMID 26478208
- [Background] Iadarola ND, Niciu MJ, Richards EM, Vande Voort JL, Ballard ED, Lundin NB, Nugent AC, Machado-Vieira R, Zarate CA Jr. Ketamine and other N-methyl-D-aspartate receptor antagonists in the treatment of depression: a perspective review. Ther Adv Chronic Dis. 2015 May;6(3):97-114. doi: 10.1177/2040622315579059. PMID 25954495
- [Background] Kavalali ET, Monteggia LM. How does ketamine elicit a rapid antidepressant response? Curr Opin Pharmacol. 2015 Feb;20:35-9. doi: 10.1016/j.coph.2014.11.005. Epub 2014 Nov 25. PMID 25462290
- [Background] Caddy C, Giaroli G, White TP, Shergill SS, Tracy DK. Ketamine as the prototype glutamatergic antidepressant: pharmacodynamic actions, and a systematic review and meta-analysis of efficacy. Ther Adv Psychopharmacol. 2014 Apr;4(2):75-99. doi: 10.1177/2045125313507739. PMID 24688759
- [Background] Lenze EJ, Farber NB, Kharasch E, Schweiger J, Yingling M, Olney J, Newcomer JW. Ninety-six hour ketamine infusion with co-administered clonidine for treatment-resistant depression: A pilot randomised controlled trial. World J Biol Psychiatry. 2016 Apr;17(3):230-8. doi: 10.3109/15622975.2016.1142607. Epub 2016 Feb 26. PMID 26919405
- [Background] Morgan CJ, Curran HV. Acute and chronic effects of ketamine upon human memory: a review. Psychopharmacology (Berl). 2006 Nov;188(4):408-24. doi: 10.1007/s00213-006-0572-3. Epub 2006 Sep 28. PMID 17006715
- [Background] Morgan CJ, Curran HV; Independent Scientific Committee on Drugs. Ketamine use: a review. Addiction. 2012 Jan;107(1):27-38. doi: 10.1111/j.1360-0443.2011.03576.x. Epub 2011 Jul 22. PMID 21777321
- [Background] Sanders RD, Weimann J, Maze M. Biologic effects of nitrous oxide: a mechanistic and toxicologic review. Anesthesiology. 2008 Oct;109(4):707-22. doi: 10.1097/ALN.0b013e3181870a17. PMID 18813051
- [Background] Nagele P, Metz LB, Crowder CM. Nitrous oxide (N(2)O) requires the N-methyl-D-aspartate receptor for its action in Caenorhabditis elegans. Proc Natl Acad Sci U S A. 2004 Jun 8;101(23):8791-6. doi: 10.1073/pnas.0402825101. Epub 2004 May 24. PMID 15159532
- [Background] Zorumski CF, Nagele P, Mennerick S, Conway CR. Treatment-Resistant Major Depression: Rationale for NMDA Receptors as Targets and Nitrous Oxide as Therapy. Front Psychiatry. 2015 Dec 9;6:172. doi: 10.3389/fpsyt.2015.00172. eCollection 2015. PMID 26696909
- [Background] Certosimo F, Walton M, Hartzell D, Farris J. Clinical evaluation of the efficacy of three nitrous oxide scavenging units during dental treatment. Gen Dent. 2002 Sep-Oct;50(5):430-5. PMID 12448895
- [Background] Myles PS, Leslie K, Chan MT, Forbes A, Peyton PJ, Paech MJ, Beattie WS, Sessler DI, Devereaux PJ, Silbert B, Schricker T, Wallace S; ANZCA Trials Group for the ENIGMA-II investigators. The safety of addition of nitrous oxide to general anaesthesia in at-risk patients having major non-cardiac surgery (ENIGMA-II): a randomised, single-blind trial. Lancet. 2014 Oct 18;384(9952):1446-54. doi: 10.1016/S0140-6736(14)60893-X. PMID 25142708
- [Background] Myles PS, Leslie K, Chan MT, Forbes A, Paech MJ, Peyton P, Silbert BS, Pascoe E; ENIGMA Trial Group. Avoidance of nitrous oxide for patients undergoing major surgery: a randomized controlled trial. Anesthesiology. 2007 Aug;107(2):221-31. doi: 10.1097/01.anes.0000270723.30772.da. PMID 17667565
- [Background] Nagele P, Brown F, Francis A, Scott MG, Gage BF, Miller JP; VINO Study Team. Influence of nitrous oxide anesthesia, B-vitamins, and MTHFR gene polymorphisms on perioperative cardiac events: the vitamins in nitrous oxide (VINO) randomized trial. Anesthesiology. 2013 Jul;119(1):19-28. doi: 10.1097/ALN.0b013e31829761e3. PMID 23856660
- [Background] Snaith RP. Present use of the Hamilton Depression Rating Scale: observation on method of assessment in research of depressive disorders. Br J Psychiatry. 1996 May;168(5):594-7. doi: 10.1192/bjp.168.5.594. PMID 8733798
- [Background] Kyle PR, Lemming OM, Timmerby N, Sondergaard S, Andreasson K, Bech P. The Validity of the Different Versions of the Hamilton Depression Scale in Separating Remission Rates of Placebo and Antidepressants in Clinical Trials of Major Depression. J Clin Psychopharmacol. 2016 Oct;36(5):453-6. doi: 10.1097/JCP.0000000000000557. PMID 27525966
- [Background] Furukawa TA, Akechi T, Azuma H, Okuyama T, Higuchi T. Evidence-based guidelines for interpretation of the Hamilton Rating Scale for Depression. J Clin Psychopharmacol. 2007 Oct;27(5):531-4. doi: 10.1097/JCP.0b013e31814f30b1. No abstract available. PMID 17873700
- [Background] Ueno F, Nakajima S, Suzuki T, Abe T, Sato Y, Mimura M, Uchida H. Whether to increase or maintain dosage of mirtazapine in early nonimprovers with depression. J Clin Psychiatry. 2015 Apr;76(4):434-9. doi: 10.4088/JCP.14m09201. PMID 25919835
- [Background] Levkovitz Y, Isserles M, Padberg F, Lisanby SH, Bystritsky A, Xia G, Tendler A, Daskalakis ZJ, Winston JL, Dannon P, Hafez HM, Reti IM, Morales OG, Schlaepfer TE, Hollander E, Berman JA, Husain MM, Sofer U, Stein A, Adler S, Deutsch L, Deutsch F, Roth Y, George MS, Zangen A. Efficacy and safety of deep transcranial magnetic stimulation for major depression: a prospective multicenter randomized controlled trial. World Psychiatry. 2015 Feb;14(1):64-73. doi: 10.1002/wps.20199. PMID 25655160
- [Background] Leucht S, Fennema H, Engel R, Kaspers-Janssen M, Lepping P, Szegedi A. What does the HAMD mean? J Affect Disord. 2013 Jun;148(2-3):243-8. doi: 10.1016/j.jad.2012.12.001. Epub 2013 Jan 26. PMID 23357658
- [Background] Gibbons RD, Weiss DJ, Pilkonis PA, Frank E, Moore T, Kim JB, Kupfer DJ. Development of a computerized adaptive test for depression. Arch Gen Psychiatry. 2012 Nov;69(11):1104-12. doi: 10.1001/archgenpsychiatry.2012.14. PMID 23117634
- [Background] Gibbons RD, Kupfer D, Frank E, Moore T, Beiser DG, Boudreaux ED. Development of a Computerized Adaptive Test Suicide Scale-The CAT-SS. J Clin Psychiatry. 2017 Nov/Dec;78(9):1376-1382. doi: 10.4088/JCP.16m10922. PMID 28493655
- [Background] Nagele P, Duma A, Kopec M, Gebara MA, Parsoei A, Walker M, Janski A, Panagopoulos VN, Cristancho P, Miller JP, Zorumski CF, Conway CR. Nitrous Oxide for Treatment-Resistant Major Depression: A Proof-of-Concept Trial. Biol Psychiatry. 2015 Jul 1;78(1):10-18. doi: 10.1016/j.biopsych.2014.11.016. Epub 2014 Dec 9. PMID 25577164
- [Background] Djulbegovic B, Hozo I, Ioannidis JP. Improving the drug development process: more not less randomized trials. JAMA. 2014 Jan 22-29;311(4):355-6. doi: 10.1001/jama.2013.283742. No abstract available. PMID 24449311